CLINICAL TRIAL: NCT05686382
Title: Anestesia Generale + TAP Block vs Anestesia Generale + CWI Per Intervento di Isterectomia Totale Laparotomica. Trial Randomizzato Controllato.
Brief Title: TAP Block vs CWI for Total Abdominal Hysterectomy, a RCT
Acronym: WI-HYSTER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Fabio Costa, Consultant Department of Anesthesia - Principal Investigator, Campus Bio-Medico University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022.178
Record Dates: First submitted 2023-01-02; First posted 2023-01-17 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group TAP block (Active Comparator): TAP block is administered at the end of the surgery, bilaterally, with lateral approach, with 24 ml of 0,5% ropivacaine for each side
  Interventions: Procedure: TAP block
- group CWI (Experimental): A 15 cm long, multihole catheter is placed on the preperitoneal plane before fascia closure; a starting bolus of 10 ml of 0,5% ropivacaine is administered through the catheter, then a continuous infusion of 0,2% ropivacaine at a rate of 5 ml/h is started through a pump and continued for 48 hours
  Interventions: Procedure: Continuous Wound Infusion

INTERVENTIONS:
Procedure: Continuous Wound Infusion — continuous local anesthetic infiltration of the wound
  Arms: group CWI
Procedure: TAP block — ultrasound guided injection of local anesthetic in the fascial plane between the internal oblique and transversus abdominis muscles
  Arms: group TAP block

SUMMARY:
This no-profit, monocentric, prospective randomized controlled trial, aims to demonstrate the non-inferiority of continuous wound infusion (CWI) when compared to transversus abdominis plane (TAP) block for postoperative pain control after total abdominal hysterectomy.

DETAILED DESCRIPTION:
After signing the informed consent, patients will be enrolled and randomly allocated into either the study group (CWI) or the control group (TAP). Both groups will receive standard general anesthesia. At the end of the surgery, the CWI patients will receive a preperitoneal catheter in the surgical wound and CWI of ropivacaine 2 mg/ml, 5 ml/h for 24 hours; with the TAP block patients will receive a bilateral, standard lateral TAP block with 5 mg/ml ropivacaine 24 ml per side. All patients will receive multimodal analgesia with ketorolac 30 mg e.v. plus 90 mg/24h IV, paracetamol 1g plus 1g TID, dexamethasone 0,1 mg/kg IV preoperatively, oxycodone 5 mg per OS upon request.

ELIGIBILITY:
Inclusion Criteria:

* ASA I - III
* laparotomic hysterectomy with Pfannenstiel incision
* signed informed consent

Exclusion Criteria:

* ASA IV
* allergy to local anesthetics or other components of multimodal analgesia
* inability to walk or eat

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 32 (Estimated)
Dates: Start 2023-01-04 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
opioid consumption | Change from baseline and hours 6, 12, 24, 48
  morphine equivalents requested (patients request oxycodone 5 mg (7,5 mg morphine equivalents) each time they experience pain at intensity higher than 4 in the NRS scale

SECONDARY OUTCOMES:
postoperative pain at rest | hours 6, 12, 24, 48
  pain at rest (numeric rating scale NRS). The patient is asked to represent her pain with a number from 0 to 10 where 0 means absence of pain and 10 means the worst pain possible
postoperative pain during movements | hours 6, 12, 24, 48
  pain at movement (numeric rating scale NRS). The patient is asked to change her position from lying to seating and represent the pain evoked by that movement with a number from 0 to 10 where 0 means absence of pain and 10 means the worst pain possible
Postoperative Nausea and Vomiting (PONV) | hours 6, 12, 24, 48
  This outcome measure would reflect a reduction in opioid consumption. One episode of PONV is registered If the patient experienced either nausea or vomiting in the specified time frame. Single episodes for any time frame and the overall number of episodes in the 48 hours are registered
early refeeding | hours 3, 12, 24, 48
  ability to drink and eat. This outcome measure would reflect a reduction in opioid consumption. The patient is asked to drink a glass of water in the specified time frame. After 10 minutes, if no nausea is experienced, the patient is asked to eat a light biscuit or similar. If tolerated, a "YES" is recorded in the specified time frame and in the subsequent ones refeeding is not investigated
early mobilization SIT-STAND-WALK | hours 3, 12, 24, 48
  Early mobilization: ability to sit, stand and walk. This outcome measure would reflect a reduction in opioid consumption and the stability of vital parameters. At the specified time frame the patient is asked to assume the sitting position. If the position change is not hampered by pain or dizziness, she is asked to stand. If the patient could stand for 10 seconds is asked to walk for 10 steps. In each time frame is recorded the kind of mobilization obtained (sit; stand; walk). After obtaining a "walk", mobility in subsequent time frames is not investigated
vital parameters stability YES/NO | hours 3, 12, 24, 48
  Mean blood pressure is measured in each time frame and compared with the baseline preoperative data. If they were found similar a "YES" is recorded. A difference from baseline > 20%. is considered to reflect poor stability and a "NO" is recorded.
vital parameter ( heart rate) stability YES/NO | hours 3, 12, 24, 48
  heart rate is measured in each time frame and compared with the baseline preoperative data. If they were found similar a "YES" is recorded. A difference from baseline > 20%. is considered to reflect poor stability and a "NO" is recorded.
vital parameter (oxygen saturation) stability YES/NO | hours 3, 12, 24, 48
  oxygen saturation are measured in each time frame and compared with the baseline preoperative data. If they were found similar a "YES" is recorded. A difference from baseline > 20%. is considered to reflect poor stability and a "NO" is recorded.
Home dischargeable YES/NO | hours 3, 12, 24, 48
  Check list for possible discharge: This outcome measure would investigate the potential for an early discharge, taking into account all the previously collected data. A check list reassuming all the outcomes will help to obtain a "YES" or a "NO" in each time frame. After obtaining a "YES", dischargeability in subsequent time frames is not investigated Check list for possible discharge: This outcome measure would investigate the potential for an early discharge, taking into account all the previously collected data. A check list reassuming all the outcomes will help to obtain a "YES" or a "NO" in each time frame. After obtaining a "YES", dischargeability in subsequent time frames is not investigated
complications | hours 0, 6, 12, 24, 48 (days 30 for DVT)
  any other possible complication is registered as description (catheter dislocation, hematoma in the TAP site, leakage from the catheter exit site, etc.) in a note in each time frame. At 30 days postoperatively, through phone interview, the patient is investigated for possible deep vein thrombosis diagnosis.
HCP time consuming | hour 0
  time needed to deliver TAP block or CWI. For each patient the time necessary to insert the catheter or to perform the TAP block is recorded
Costs of all procedure | hour 0
  difference in costs between groups. Costs of all procedure related costs are taken into account (drugs, devices, HCP time, OR time) and compared

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Costa, Dr., Principal Investigator — Fondazione Policlinico Universitario Campus Biomedico di Roma
Locations (1):
- CampusBioMedico, Rome, Italy